CLINICAL TRIAL: NCT00320307
Title: An Open-Label, Two-Period, Crossover, Pharmacokinetic Study of Abacavir and Its Intracellular Anabolite Carbovir Triphosphate Following Once-Daily and Twice-Daily Administration of Abacavir in HIV-Infected Subjects.
Brief Title: Comparison of Abacavir Following Once-Daily And Twice-Daily Administration In HIV Infected Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CAL102120
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: HIV Infection
Keywords: Human Immunodeficiency Virus; HIV; Abacavir regime; ABC
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — abacavir

INTERVENTIONS:
Drug: abacavir

SUMMARY:
The purpose of the study is to look at the levels of the drug abacavir (ABC) in blood. Also, the study will look at the levels of carbovir triphosphate (CBV-TP), which is the active substance produced from ABC in the bodyâ s cells which helps prevent HIV from multiplying. CBV-TP will be measured in specific blood cells. The amount of ABC and CBV-TP will be looked at when subjects receive ABC as a 300mg dose twice a day and compared with the levels when they receive ABC as a 600mg dose once a day.

ELIGIBILITY:
Inclusion criteria:

* Healthy adults , inclusively.
* Documented HIV-1 infection (documented by historical data or current validated assay).
* Undetectable viral load.
* Currently on an ABC-tablet containing regimen for at least 8 weeks.
* Willingness to temporarily switch ABC schedule from BID to QD, or vice versa, for 11 days.
* Weigh between 40-100kg, inclusive.

Exclusion criteria:

* Subjects who are receiving tenofovir.
* Previous study participation in other experimental drug trial(s) within 30 days before the screening phase of the study.
* Subjects who currently regularly take drugs-of-abuse, with the exception of cannabinoids.
* Subjects who cannot refrain from taking herbal remedies during the course of the study.
* Subjects who regularly consume more than an average amount of alcohol per day.
* Poor general health preventing fasting or blood sampling.
* Subjects who are not able to discontinue use of hydroxyurea, mycophenolate or ribavirin for 14 days prior to entering the study until discharge from the study.
* An unwillingness of a male subject to abstain from sexual intercourse with women of childbearing potential or an unwillingness to use a condom in addition to having their female partner use another form of contraception.
* The subject is pregnant or nursing an infant.
* History of symptoms consistent with a hypersensitivity reaction to ABC.
* Positive HCV Antibody or HepBsAg (Hepatitis B surface antigen).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-09

PRIMARY OUTCOMES:
To assess the pharmacokinetics of intracellular CBV-TP at steady state following administration of 600 mg QD and 300 mg BID ABC-containing regimens in HIV infected adult subjects. | throughout the study

SECONDARY OUTCOMES:
- To compare plasma concentrations of ABC, and intracellular CBV-TP - To assess the safety and tolerability of dosing with ABC 300mg BID and 600mg QD. - To assess potential gender effects in the pharmacokinetics of ABC. | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom